CLINICAL TRIAL: NCT01254916
Title: The Sinonasal Outcome Test - 22, Validated for Danish Patients
Status: Completed | Type: Observational
Sponsor: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Bibi Lange, MD, Ph.d.-student, Odense University Hospital
Other Study IDs: Danish SNOT 22
Record Dates: First submitted 2010-12-06; First posted 2010-12-07 (Estimated); Last update posted 2012-05-08 (Estimated); Status verified 2012-05

CONDITIONS: Chronic Rhinosinusitis
Keywords: Chronic Rhinosinusitis; Sinonasal Outcome test 22

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Patients with chronic rhinosinusitis

SUMMARY:
Introduction: Chronic rhinosinusitis (CRS) is a significant health problem increasing in both incidence and prevalence. It calls into attention consensus about diagnosing, assessing symptoms and treatment of patients with CRS. Therefore a validated Danish measure of health-related quality of life in sinonasal disease is needed.

Method: The Sinonasal Outcome measure 22 (SNOT-22) was translated into Danish and reproducibility was evaluated by test-retesting 40 patients with CRS. The statistical analyses used, were Pearson´s correlation coefficient, Cronbach´s alfa, Kappa and Bland-Altman´s Plot. Reproducibility was also tested looking at subscales within the SNOT-22.

Result: The results show good internal correlation with Cronbach´s alfa at 0.83 in the initial test and 0.92 in the retest. Pearson was 0.70 (p<0.001) revealing good correlation between the initial scores and the retests scores. Kappa was calculated for each item with a mean value of 0.61 showing substantial agreement. Paired t-test revealed no significant difference in the subscales.

Conclusion: The Danish version of SNOT-22 is recommended for Danish clinicians and researches as a patient-reported measure of outcome in sino-nasal disorders such as rhinosinusitis and nasal polyposis.

ELIGIBILITY:
Inclusion Criteria: Persons diagnosed with Chronic Rhinosinusitis -

Exclusion Criteria: Change of treatment or acute change of symptoms due to common cold/influenza in the time between completing the test and the retest. If SNOT-score was very low. Persons who left before offered test or declined testing.

-

Ages: 15 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with chronic rhinosinusitis diagnosed by a medical doctor
Sampling Method: Non-Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2008-10; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Reproducibility of Sinonasal Outcome test 22 | From the time of fullfilling the first SNOT-22 to fullfilling the second SNOT-22 after 14 days

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Otorhinolaryngology, Odense University Hopsital, Odense, Denmark

REFERENCES:
- [Derived] Lange B, Thilsing T, Al-kalemji A, Baelum J, Martinussen T, Kjeldsen A. The Sino-Nasal Outcome Test 22 validated for Danish patients. Dan Med Bull. 2011 Feb;58(2):A4235. PMID 21299922